CLINICAL TRIAL: NCT02769403
Title: Using a Daily Mindfulness Practice With Biofeedback to Improve Job Satisfaction and Performance in a Primary Care Outpatient Clinic
Brief Title: Mindfulness With Biofeedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 201600018
Record Dates: First submitted 2016-04-22; First posted 2016-05-11 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2017-05

CONDITIONS: Mindfulness Training
Keywords: Job Satisfaction; Job Performance; Primary Care
MeSH Terms: interventions — Surveys and Questionnaires; Blood Pressure; Heart Rate; Sick Leave

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants will use HeartMath EmWave Pro for at least one 5-minute session daily, Monday through Friday. The treatment participants will use it daily for all 12 weeks, and will have the added component of weekly visits for the first 6 weeks of the study from the study team. The weekly visits is focused on reinforcing accountability and achievement of coherence. The participants will also complete questionnaires at baseline, week 6, and week 12 about demographics, job satisfaction, and job performance. Participants' blood pressure and heart rate will be collected at those three time points. Additionally, information about participants' use of HeartMath EmWave Pro, sick days, and patient satisfaction will be collected after week 12.
  Interventions: Device: HeartMath EmWAVE Pro; Other: Questionnaires; Other: Blood Pressure and Heart Rate; Other: Sick Days; Other: Patient Satisfaction
- Control (Active Comparator): Participants will use HeartMath EmWave Pro for at least one 5-minute session daily, Monday through Friday. The control participants will use it daily only for weeks 7-12. The participants will also complete questionnaires at baseline, week 6, and week 12 about demographics, job satisfaction, and job performance. Participants' blood pressure and heart rate will be collected at those three time points. Additionally, information about participants' use of HeartMath EmWave Pro, sick days, and patient satisfaction will be collected after week 12.
  Interventions: Device: HeartMath EmWAVE Pro; Other: Questionnaires; Other: Blood Pressure and Heart Rate; Other: Sick Days; Other: Patient Satisfaction

INTERVENTIONS:
Device: HeartMath EmWAVE Pro — The following information will be recorded about HeartMath use:
  Self-report: adherence (whether the daily session was completed), coherence score, any comments/notes about the daily session From the application: coherence ratio, coherence score, achievement score, session time, average heart rate
Other: Questionnaires — All participants will complete questionnaires at baseline, week 6, and week 12 about demographics, job satisfaction, and job performance.
Other: Blood Pressure and Heart Rate — All participants will have blood pressure and heart rate collected at baseline, week 6, and week 12.
Other: Sick Days — Sick days during the 12 week study period will be collected
Other: Patient Satisfaction — This will include patients who complete the satisfaction survey for the 12 weeks prior to the study and during the 12 week study period. Each patient satisfaction survey is tied to a specific healthcare provider (physicians, Advanced Registered Nurse Practitioner (ARNP) & Physician Assistants [advance practice clinicians], and nurses) and will be linked to the consented research participant.

SUMMARY:
The purpose of this research study is to determine if using HeartMath's biofeedback with emWave Pro daily mindfulness practice: is a practical and effective intervention to improve job satisfaction and performance of physicians, advance practice clinicians, and nurses; improves patient satisfaction; and affects resting blood pressure and heart rate when comparing baseline to follow-up measures.

DETAILED DESCRIPTION:
This research study seeks to determine if using a daily mindfulness practice with EmWave Pro HeartMath helps to achieve coherence through various standardized, interactive mindfulness techniques, such as guided meditations focusing on positive emotions, breathing, and imagery. The investigators seek to determine if using HeartMath's biofeedback with emWave Pro daily mindfulness practice: is a practical and effective intervention to improve job satisfaction and performance of physicians, advance practice clinicians, and nurses; improves patient satisfaction; and affects resting blood pressure and heart rate when comparing baseline to follow-up measures.

All participants will attend a one-time one-hour training session to explain cardiac coherence and how to use emWave Pro. Participants will be randomized to be either in the treatment group or the control group. Participants will use emWave Pro for at least one 5-minute session daily, Monday through Friday. The treatment participants will use it daily for all 12 weeks. The control participants will use it daily only for weeks 7-12. The treatment group will have the added component of weekly visits during the first 6 weeks of the study from an investigator and the research coordinator. The purpose of the weekly visits is focused on reinforcing accountability and achievement of coherence.

The participants will also complete questionnaires at baseline, week 6, and week 12 about demographics, job satisfaction, and job performance. Participants' blood pressure and heart rate will be collected at those three time points. Additionally, information about participants' use of HeartMath, sick days, and patient satisfaction will be collected after week 12.

ELIGIBILITY:
Inclusion Criteria:

* Individuals (physicians, Advanced Registered Nurse Practitioner (ARNPs) & Physician Assistants [advance practice clinicians], and nurses) working at the two research sites: Hampton Oaks and Haile Plantation at UF Health

Exclusion Criteria:

* Anyone not working at Hampton Oaks and Haile Plantation at UF Health

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-06; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Changes in Minnesota Satisfaction Questionnaire - Short Form will be used to determine job satisfaction at baseline, week 6, and week 12 | Change from baseline, week 6, and week 12
  The Minnesota Satisfaction Questionnaire - Short Form (MSQ-SF) uses a 5-point Likert-type scale with 20 items. Responses range from 1 (very satisfied) - 5 (very dissatisfied) so the lower the score the higher the job satisfaction and the higher the score the lower the job satisfaction.
Changes in Perceived Stress Scale will be used to determine job satisfaction at baseline, week 6, and week 12 | Change from baseline, week 6, and week 12
  The Perceived Stress Scale (PSS) has a range of scores between 0 and 40. A higher score indicates more stress.
Changes in Medical Office Survey on Patient Safety will be used to determine job performance between at baseline, week 6, and week 12 | Change from baseline, week 6, and week 12
  The Medical Office Survey on Patient Safety (MOSOPS) is a 51-item survey that measures 12 domains of office culture conceptually related to patient safety. The lower the overall score the less job performance and the higher the score the better the job performance.
The number of sick days will be assessed | During 12 week period

SECONDARY OUTCOMES:
Changes in blood pressure between the groups from baseline, week 6, and week 12 | Change from baseline, week 6, and week 12
Changes in heart rate between the groups from baseline, week 6, and week 12 | Change from baseline, week 6, and week 12
UF Physicians Faculty (UFP) Practice: Patient Satisfaction Survey | For the 12 weeks prior to the study and during the 12 week study period
  The patient satisfaction surveys are used by clinics in the UF Physicians Faculty (UFP) Practice and are managed by UFP administration. Patients are asked questions about rating their visit, instructions and explanations given during the visit, appointment scheduling, wait time, customer service, and demographics.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Orlando, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Hampton Oaks, Gainesville, Florida
  - Halie Plantation, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Undecided